CLINICAL TRIAL: NCT05706623
Title: A Phase 1, Open-Label Evaluation of the Pharmacokinetics and Safety of a Single Dose of Apraglutide in Subjects With Normal and Impaired Hepatic Function
Brief Title: A Phase 1 Open-Label Evaluation of the Pharmacokinetics and Safety of a Single Dose of Apraglutide in Subjects With Normal and Impaired Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VectivBio AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TA799-015
Record Dates: First submitted 2023-01-20; First posted 2023-01-31 (Actual); Results first posted 2025-06-13 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-06

CONDITIONS: Hepatic Impairment
Keywords: Hepatic Impairment; Liver Function; Hepatic Function
MeSH Terms: interventions — apraglutide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: Moderate hepatic impairment (Experimental): Child-Pugh B
  Interventions: Drug: Apraglutide
- Part 1: Normal hepatic function (Experimental)
  Interventions: Drug: Apraglutide
- Part 2: Mild hepatic impairment (Experimental): Child-Pugh A
  Interventions: Drug: Apraglutide

INTERVENTIONS:
Drug: Apraglutide — Single dose of apraglutide

SUMMARY:
The primary objective is to assess the pharmacokinetics (PK) of apraglutide in subjects with hepatic impairment compared with matched control subjects with normal hepatic function following single subcutaneous (SC) dose administration.

DETAILED DESCRIPTION:
A two stage design, open label, multi-center, non-randomized trial to evaluate the the safety and tolerability of a single subcutaneous dose of apraglutide in subjects with varying degrees of hepatic function. The hepatic function will estimated with the Child-Pugh classification.

Part 1: 8 subjects with moderate hepatic impairment (Cohort 1) and 8 subjects with normal hepatic function (Cohort 2).

Part 2: 8 subjects with mild hepatic impairment (Cohort 3) and 8 subjects with normal hepatic function (from Cohort 2 where possible and additional subject). Part 2 will be conducted only if the geometric mean ratio (GMR) of area under the curve extrapolated to infinity (AUCinf) or area under the curve from zero to the last measurable point (AUClast) for the moderate hepatic impairment group compared to the control group is ≥2.

ELIGIBILITY:
Inclusion Criteria:

All Participants:

* Age between 18 and 75 years inclusive
* Subjects who are willing and able to comply with the study procedures
* Subjects able to understand and willing to sign the informed consent
* Body mass index (BMI) of ≥18 to ≤35 kg/m2; and a total body weight of >50 kg (110 lb).
* Women of childbearing potential (WOCBP) on highly effective method of contraception during the trial and for 1 month after the end of trial (EOT) visit. Sterilized or infertile or postmenopausal females.
* Male subjects with a female partner of childbearing potential: highly effective methods of contraception and no sperm donation during the trial and for 1 month after (EOT) visit.

Participants with impaired hepatic function:

* Confirmed and documented diagnosis of cirrhosis
* Moderate liver disease (Child-Pugh B): clinically stable for at least 1 month prior to screening
* Mild liver disease (Child-Pugh A): clinically stable for at least 1 month prior to screening

Exclusion Criteria:

* History of clinically significant GI, bronchopulmonary, neurological, cardiovascular, endocrine, or allergic disease
* Known hypersensitivity to the investigational medicinal product (IMP), any of their excipients or drugs of the same class
* If capable of reproduction, unwilling to use an effective form of contraception
* If a female of child-bearing potential, a positive urine/blood pregnancy test
* Breast-feeding women
* Positive urine/blood test for alcohol and drugs of abuse at Screening and on Day-1
* Use of prohibited medications or herbal remedies
* Known presence or history of intestinal polyps
* Known presence or history of any type of cancer
* Pancreatic events such as acute pancreatitis, pancreatic duct stenosis, pancreas infection, and increased blood amylase and lipase (>2.0-5.0×upper limit of normal range)
* Participation in an investigational drug or device study within 30 days prior to Screening
* Donation of blood over 500 mL within 2 months prior to Screening
* Heavy use of tobacco products (i.e., smokes more than 10 cigarettes per day)
* Concomitant disease or condition that could interfere with, or for which the treatment of might interfere with, the conduct of the study, or that would, in the opinion of the Investigator, pose an unacceptable risk to the subject in this trial
* Any intercurrent clinically significant illness in the previous 28 days before Day 1 of this study
* Positive blood screen for human immunodeficiency virus (HIV) antigen/antibody combo, hepatitis A (HAV), hepatitis B surface antigen (HBsAgB), or hepatitis C virus (HCV)
* Unwillingness or inability to comply with the study protocol for any other reason

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2023-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Masior, Study Director — VectivBio AG
Locations (2):
- APEX, Münich, Germany
- Summit Clinical Research, Bratislava, Slovakia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in 2 study sites in Slovakia and Germany and participated from February 2023 to April 2023.
Pre-assignment Details: In Part 1, participants with normal hepatic function were matched 1:1 for age (±10 years), body mass index (BMI; ±15%), and sex (1:1) to participants with moderate hepatic impairment. Part 2 was to be conducted dependent on the outcome of Part 1 and planned to enroll participants with mild hepatic impairment. No participants enrolled in Part 2.
Groups:
- Normal Hepatic Function Group: Participants with normal hepatic function received a single subcutaneous (SC) dose of apraglutide on Day 1.
- Moderate Hepatic Impairment Group: Participants with moderate hepatic impairment received a single SC dose of apraglutide on Day 1.
Period: Overall Study
Arm/Group | Normal Hepatic Function Group | Moderate Hepatic Impairment Group
Started | 8 | 8
Dosed With Apraglutide | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Normal Hepatic Function Group: Participants with normal hepatic function received a single SC dose of apraglutide on Day 1.
- Total: Total of all reporting groups
Arm/Group | Normal Hepatic Function Group | Moderate Hepatic Impairment Group | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Full Range); unit: years] | 58.3 [41 to 71] | 58.8 [42 to 75] | 58.5 [41 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 5 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 8 | 16
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 8 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve to Infinity (AUCinf) of Apraglutide
Description: Apraglutide was quantified in human plasma samples using a fully validated liquid chromatography mass spectrometry-based method, with a lower limit of quantification (LLOQ) of 1 ng/mL and an upper limit of 200 ng/mL. Plasma pharmacokinetic (PK) parameters for apraglutide were estimated using non-compartmental methods from the concentration-time profiles. Actual sampling times, rather than scheduled sampling times, were used. AUCinf was calculated as: AUCinf = AUC from time zero to the last quantifiable concentration (AUClast) + (Clast/kel) where Clast was the observed concentration at the last time point with concentrations above the lower limit of quantification and kel was the terminal elimination rate constant.
Time Frame: Pre-dose Day 1; 6, 12, 24, 28, 36, 40, 48, 60, 72, 96, 120, 144, 168, 240, and 312 hours post-dose
Population: The PK parameter set included participants who received at least one dose of apraglutide and who had at least one PK parameter of interest estimated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Normal Hepatic Function Group | Moderate Hepatic Impairment Group
Number analyzed (Participants) | 8 | 8
h*ng/mL | 4481 (64.5) | 3744 (50.2)
Statistical Analysis 1: Comparison: Normal Hepatic Function Group vs Moderate Hepatic Impairment Group; Moderate Hepatic Impairment Group (test) versus Normal Hepatic Function Group (reference). The analysis was performed on natural log (ln) transformed parameters using an analysis of variance model with the hepatic function group as a fixed effect; Test type: Other — Analysis of variance model; Geometric least squares (LS) mean ratio = 0.8354, 90% CI 2-sided [0.5216 to 1.338]

2. Primary Outcome: Area Under the Curve (AUC) From Time Zero to 168 Hours Post-dose (AUC0-168h) of Apraglutide
Description: Apraglutide was quantified in human plasma samples using a fully validated liquid chromatography mass spectrometry-based method, with a LLOQ of 1 ng/mL and an upper limit of 200 ng/mL. Plasma PK parameters for apraglutide were estimated using non-compartmental methods from the concentration-time profiles. Actual sampling times, rather than scheduled sampling times, were used.
Time Frame: Pre-dose Day 1; 6, 12, 24, 28, 36, 40, 48, 60, 72, 96, 120, 144, and 168 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Normal Hepatic Function Group | Moderate Hepatic Impairment Group
Number analyzed (Participants) | 8 | 8
h*ng/mL | 4271 (65.2) | 3605 (50.2)

3. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Apraglutide
Description: Apraglutide was quantified in human plasma samples using a fully validated liquid chromatography mass spectrometry-based method, with a LLOQ of 1 ng/mL and an upper limit of 200 ng/mL. Plasma PK parameters for apraglutide were estimated using non-compartmental methods from the concentration-time profiles. Actual sampling times, rather than scheduled sampling times, were used. Cmax was the observed peak analyte concentration obtained directly from the experimental data without interpolation, expressed in concentration units.
Time Frame: Pre-dose Day 1; 6, 12, 24, 28, 36, 40, 48, 60, 72, 96, 120, 144, 168, 240, and 312 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Normal Hepatic Function Group | Moderate Hepatic Impairment Group
Number analyzed (Participants) | 8 | 8
ng/mL | 58.3 (68.3) | 54.6 (43.1)
Statistical Analysis 1: Comparison: Normal Hepatic Function Group vs Moderate Hepatic Impairment Group; Moderate Hepatic Impairment Group (test) versus Normal Hepatic Function Group (reference). The analysis was performed on ln transformed parameters using an analysis of variance model with the hepatic function group as a fixed effect; Test type: Other — Analysis of variance model; Geometric LS Mean Ratio = 0.9356, 90% CI 2-sided [0.5889 to 1.4864]

4. Secondary Outcome: Time of Maximum Plasma Concentration (Tmax) of Apraglutide
Description: Apraglutide was quantified in human plasma samples using a fully validated liquid chromatography mass spectrometry-based method, with a LLOQ of 1 ng/mL and an upper limit of 200 ng/mL. Plasma PK parameters for apraglutide were estimated using non-compartmental methods from the concentration-time profiles. Actual sampling times, rather than scheduled sampling times, were used. Tmax was the first observed time to reach peak analyte concentration obtained directly from the experimental data without interpolation, expressed in time units.
Time Frame: Pre-dose Day 1; 6, 12, 24, 28, 36, 40, 48, 60, 72, 96, 120, 144, 168, 240, and 312 hours post-dose
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Normal Hepatic Function Group | Moderate Hepatic Impairment Group
Number analyzed (Participants) | 8 | 8
hours | 32.03 [27.97 to 48.15] | 31.76 [12.00 to 36.00]

5. Secondary Outcome: Apparent Clearance After Extravascular Administration (CL/F) of Apraglutide
Description: as for outcome 2
Time Frame: Pre-dose Day 1; 6, 12, 24, 28, 36, 40, 48, 60, 72, 96, 120, 144, 168, 240, and 312 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Normal Hepatic Function Group | Moderate Hepatic Impairment Group
Number analyzed (Participants) | 8 | 8
L/h | 1.12 (64.5) | 1.34 (50.2)

6. Secondary Outcome: Terminal Elimination Rate Constant (Kel) of Apraglutide
Description: Apraglutide was quantified in human plasma samples using a fully validated liquid chromatography mass spectrometry-based method, with a LLOQ of 1 ng/mL and an upper limit of 200 ng/mL. Plasma PK parameters for apraglutide were estimated using non-compartmental methods from the concentration-time profiles. Actual sampling times, rather than scheduled sampling times, were used. Terminal elimination rate constant calculated by linear regression of the terminal log-linear portion of the concentration vs. time curve. Linear regression of at least three points and an adjusted r^2 greater than or equal to 0.80 were required to obtain a reliable kel.
Time Frame: Pre-dose Day 1; 6, 12, 24, 28, 36, 40, 48, 60, 72, 96, 120, 144, 168, 240, and 312 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/h
Arm/Group | Normal Hepatic Function Group | Moderate Hepatic Impairment Group
Number analyzed (Participants) | 8 | 8
1/h | 0.0209 (51.6) | 0.0237 (44.4)

7. Secondary Outcome: Terminal Half-life (t1/2) of Apraglutide
Description: as for outcome 2
Time Frame: Pre-dose Day 1; 6, 12, 24, 28, 36, 40, 48, 60, 72, 96, 120, 144, 168, 240, and 312 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Normal Hepatic Function Group | Moderate Hepatic Impairment Group
Number analyzed (Participants) | 8 | 8
hours | 33.2 (51.6) | 29.2 (44.4)

8. Secondary Outcome: Apparent Volume of Distribution After Extravascular Administration (Vz/F) of Apraglutide
Description: as for outcome 2
Time Frame: Pre-dose Day 1; 6, 12, 24, 28, 36, 40, 48, 60, 72, 96, 120, 144, 168, 240, and 312 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Normal Hepatic Function Group | Moderate Hepatic Impairment Group
Number analyzed (Participants) | 8 | 8
liters | 53.4 (91.1) | 56.2 (69.4)

9. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: A TEAE was any unfavorable and unintended sign, symptom, or disease temporally associated with apraglutide, whether or not related, that occurred or worsened after the dose of apraglutide. A serious TEAE was defined as any TEAE that resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect or was an important medical event. TEAEs were graded for severity based on the National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0 as follows from Grade 1 (mild) to Grade 5 (AE resulted in death). Clinically significant changes in physical examination findings, laboratory results, vital signs, and 12-lead electrocardiograms (ECGs) were also recorded as TEAEs.
Time Frame: Day 1 to Day 14
Population: The safety analysis set included all participants who received at least one dose of apraglutide.
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Hepatic Function Group | Moderate Hepatic Impairment Group
Number analyzed (Participants) | 8 | 8
Participants
  At least one TEAE | 0 | 1
  At least one serious TEAE | 0 | 0
  At least one TEAE leading to discontinuation | 0 | 0
  Any mild TEAE | 0 | 1
  Any moderate TEAE | 0 | 1
  Any related TEAE | 0 | 1

ADVERSE EVENTS:
Time Frame: Day 1 to Day 14
Description: The safety analysis set included all participants who received at least one dose of apraglutide.
Arm/Group | Normal Hepatic Function Group | Moderate Hepatic Impairment Group
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 1/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Normal Hepatic Function Group (N=8) | Moderate Hepatic Impairment Group (N=8)
Headache (Nervous system disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Part 2 was to be conducted if the geometric mean ratio (GMR) point estimate of apraglutide AUCinf or AUClast for the moderate hepatic impairment group compared with the control group was ≥2. As the GMR point estimate of AUCinf was <2, the trial stopped after Part 1.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-10-06): https://cdn.clinicaltrials.gov/large-docs/23/NCT05706623/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-03): https://cdn.clinicaltrials.gov/large-docs/23/NCT05706623/SAP_001.pdf